CLINICAL TRIAL: NCT01918085
Title: Open, Prospective, Single Centre, Randomized, Controlled, Cross-over. Clinical Study Investigating the Correlation in Peel Force of Standard Hydrocolloid Adhesive and a Standard Strata Adhesive From Peristomal Skin and Pre-stripped Abdominal Skin in Colostomists
Brief Title: Human Skin Test Model in Colostomists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CP228
Record Dates: First submitted 2013-08-06; First posted 2013-08-07 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2014-01

CONDITIONS: Colostomy Stoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peristomal skin (Other): The peel force used to remove two types of adhesive strips (Hydrocolloid strip and strata strip) from the Peristomal skin
  Interventions: Other: Hydrocolloid strip; Other: Strata strip
- Pre-stripped abdominal skin (Other): The peel force used to remove two types of adhesive strips (Hydrocolloid strip and strata strip) from healthy abdominal skin
  Interventions: Other: Hydrocolloid strip; Other: Strata strip

INTERVENTIONS:
Other: Hydrocolloid strip — An adhesive strip made of hydrocolloid adhesive
Other: Strata strip — An adhesive strip made of the Strata adhesive

SUMMARY:
The aim of the study is to investigate the correlation in peel force when peeling off a standard hydrocolloid adhesive strip and standard strata adhesive strip from peristomal skin compared to pre-stripped healthy abdominal skin in colostomists.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent.
2. Be in the age of 45 to 75 years of age both extremes included.
3. Have had a colostomy for at least 1 year.
4. Has a colostomy with a diameter up to (≤) 40 mm.
5. Have mental capacity to understand the study guidelines and questionnaires.
6. Be assessed by the investigator as having a peristomal and abdominal skin condition justifying entry into the investigation.
7. Are colostomists currently using a 1-piece and 2-piece flat ostomy appliance.
8. Have a BMI between 20-30 kg/m2.
9. Are willing to comply with investigation procedures.

Exclusion Criteria:

1. Currently suffering from peristomal skin problems (i.e. bleeding or broken skin).
2. Received radio- and/or chemotherapy within the last two months.
3. Currently using or have within the last 3 weeks used topical steroid products or other skin prep products.

   on peristomal skin (injections and oral treatment are accepted).
4. Have dermatological problems.
5. Participating in other clinical studies or have previously participated in this test.
6. Be a daily user of a convex base-plate.
7. Are pregnant or breastfeeding.
8. Systemic elements that could affect skin histology (e.g. liver, kidney or immunological diseases).

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tonny Karlsmark, MD, Principal Investigator — Bispebjerg Hospital, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited in April 2012.All subjects were recruited to one site. Copenhagen Wound Healing Centre, Bispebjerg bakke 23, 2400 Copenhagen NV Denmark.
Pre-assignment Details: Subjects must have an colostomy under 40 mm in Diameter. One subject was not randomised as the subject had a stoma with a diameter above 40 mm.
  Thus, 22 subjects were randomized.
Groups:
- First Pre-stripped Abdominal Skin, Then Peristomal Skin: The peel force used to remove two types of adhesive strips (Hydrocolloid strip and strata strip) from healthy abdominal skin
  Strata strip : An adhesive strip made of the Strata adhesive
  Hydrocolloid strip : An adhesive strip made of hydrocolloid adhesive
- First Peristomal Skin, Then Pre-stripped Abdomianl Skin: The peel force used to remove two types of adhesive strips (Hydrocolloid strip and strata strip) from the Peristomal skin
  Strata strip : An adhesive strip made of the Strata adhesive
  Hydrocolloid strip : An adhesive strip made of hydrocolloid adhesive
Period: Test Period 1: Strata Strip
Arm/Group | First Pre-stripped Abdominal Skin, Then Peristomal Skin | First Peristomal Skin, Then Pre-stripped Abdomianl Skin
Started | 10 | 12
Completed | 10 | 11
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Test Period 1: Hydrocolloid Strip
Arm/Group | First Pre-stripped Abdominal Skin, Then Peristomal Skin | First Peristomal Skin, Then Pre-stripped Abdomianl Skin
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0
Period: Test Period 2: Strata Strip
Arm/Group | First Pre-stripped Abdominal Skin, Then Peristomal Skin | First Peristomal Skin, Then Pre-stripped Abdomianl Skin
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0
Period: Test Period 2: Hydrocolloid Strip
Arm/Group | First Pre-stripped Abdominal Skin, Then Peristomal Skin | First Peristomal Skin, Then Pre-stripped Abdomianl Skin
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Pre-stripped Abdominal Skin: The peel force used to remove two types of adhesive strips (Hydrocolloid strip and strata strip) from healthy abdominal skin
  Strata strip : An adhesive strip made of the Strata adhesive
  Hydrocolloid strip : An adhesive strip made of hydrocolloid adhesive
- Peristomal Skin: The peel force used to remove two types of adhesive strips (Hydrocolloid strip and strata strip) from the Peristomal skin
  Strata strip : An adhesive strip made of the Strata adhesive
  Hydrocolloid strip : An adhesive strip made of hydrocolloid adhesive
- Total: Total of all reporting groups
Arm/Group | Pre-stripped Abdominal Skin | Peristomal Skin | Total
Number analyzed (Participants) | 10 | 12 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (5.8) | 63.5 (7.9) | 64.4 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Peel Force
Description: The peel force was measured with a tensile tester which measured the force needed to remove the the adhesive strip from the skin with a constant speed 304mm/min and a mean angel of 90 degrees.
  The peel force was measured on all participants in the flow module. However, sometimes the measurements failed and therefore did not provide a result. In example a wheel chair user was included and non of peel force measurements were succesful on the subject. The rest of the failed measurements were distributed randomly between the subjects.
Time Frame: 1 hour
Population: Some of the measurements failed. i.e one subject was a wheel chair user and the peel force could not be measured on this person.
  Only the measurements that did not fail were included in the analysis
Measure: Mean (Standard Deviation); unit: Newton
Groups:
- Peristomal Skin- Strata Adhesive: The peel force used to remove a strata strip) from the Peristomal skin
  Strata strip : An adhesive strip made of the Strata adhesive
- Pre-stripped Abdominal Skin -Strata Adhesive: The peel force used to remove a strata strip from healthy abdominal skin
  Strata strip : An adhesive strip made of the Strata adhesive
- Pre-stripped Abdominal Skin - Hydrocolloid Adhesive; Peristomal Skin - Hydrocolloid Adhesive: The peel force used to remove a hydrocolloid strip from the Peristomal skin
  hydrocolloid strip : An adhesive strip made of the hydrocolloid adhesive
Arm/Group | Peristomal Skin- Strata Adhesive | Pre-stripped Abdominal Skin -Strata Adhesive | Pre-stripped Abdominal Skin - Hydrocolloid Adhesive | Peristomal Skin - Hydrocolloid Adhesive
Number analyzed (Participants) | 19 | 18 | 19 | 20
Newton | 2.6 (1.1) | 2.1 (0.8) | 4.4 (1.8) | 3.4 (1.4)

ADVERSE EVENTS:
Arm/Group | Pre-stripped Abdominal Skin | Peristomal Skin
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 1/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre-stripped Abdominal Skin (N=22) | Peristomal Skin (N=22)
Itching related to a gall stone incident (Hepatobiliary disorders) | 0 (0) | 1 (1) — Not related to the investigational device
Pain related to a gall stone incident (Hepatobiliary disorders) | 0 (0) | 1 (1) — not related to the investigational device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No